CLINICAL TRIAL: NCT02419196
Title: Perioperative Change of Regional Ventilation During Spontaneous Breathing
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: perioperativeEIT
Record Dates: First submitted 2014-12-01; First posted 2015-04-17 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Pulmonary Infection; Pleural Effusion; Atelectasis; Pneumothorax; Bronchospasm; Aspiration Pneumonitis; Respiratory Insufficiency
MeSH Terms: conditions — Pleural Effusion; Pulmonary Atelectasis; Pneumothorax; Bronchial Spasm; Pneumonia, Aspiration; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- abdominal surgery: 27 patients undergoing abdominal surgery having an elevated risk for postoperative pulmonary complications will be examined by perioperative pulmonary function tests
  Interventions: Other: Perioperative pulmonary function tests
- limb surgery: 27 patients undergoing upper and lower limb surgery having an elevated risk for postoperative pulmonary complications will be examined by perioperative pulmonary function tests
  Interventions: Other: Perioperative pulmonary function tests
- flail chest: 10 patients undergoing an operative stabilization of a flail chest will be examined by perioperative pulmonary function tests
  Interventions: Other: Perioperative pulmonary function tests

INTERVENTIONS:
Other: Perioperative pulmonary function tests — Pulmonary electrical impedance tomography, spirometry, pulse oximetry and query performed preoperatively, at the first and the third postoperative day

SUMMARY:
Perioperative changes in regional ventilation by pulmonary electrical impedance tomography and spirometry will be investigated in patients at risk for postoperative pulmonary complications. Those patients undergo abdominal and limb operations. In a pilot study arm electrical impedance tomography is tested in patients receiving osteosynthesis of serial rib fractures.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (Defined as pulmonary infection, pleural effusion, atelectasis, pneumothorax, bronchospasm, aspiration pneumonitis or respiratory insufficiency subsequent to surgery) increase the morbidity and mortality of surgical patients. Several independent factors determined by the patients' characteristics and the operative procedure increase the risk for those complications. The postoperative decrease of values measured by spirometry, such as the forced vital capacity (FVC) and forced expiratory volume in one second (FEV1), were found in patients after major surgical procedures for several days. The postoperative reduction of those measurement can be the result of general functional limitations in those patients (e.g. by postoperative pain) or the result of a regional postoperative pulmonary complication (e.g. atelectasis, pleural effusion). The method of the electrical impedance tomography (EIT) enables to visualize the regional ventilation within a transversal section of the lung in real time. Studies examining the change of pulmonary EIT for several days postoperatively in spontaneously breathing patients are lacking. The aim of the present study is to examine perioperative changes in regional ventilation in spontaneously breathing patients during their recovery after abdominal and limb surgery. Moreover, the association of those changes with expected changes in spirometry is tested. Finally, in patients with evident postoperative pulmonary complications the value of pulmonary EIT to detect those changes is investigated. The study should improve the knowledge about the development of postoperative pulmonary complications and test the scientific and clinical value of pulmonary EIT in those spontaneously breathing patients.

In a group of patients undergoing osteosynthesis of a flail chest, it is tested how regional ventilation changes by these operations and whether pulmonary EIT is actually usable in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Inpatient
* Surgery under general anesthesia with and without additional regional anesthesia
* increased risk for postoperative pulmonary complications according to the ARISCAT-Score (except pilot arm for osteosynthesis of flail chest)

Exclusion Criteria:

* Missing informed consent
* Outpatient
* Emergency procedure
* Revision surgery of hospitalized patients
* Operation under local or regional anesthesia alone
* Expected postoperative ventilation
* Expected hospital stay of less than three days
* Pregnancy
* Allergy against material of the electrode belt (silicone rubber, stainless steel, gold-plated brass)
* Injured, inflamed or otherwise affected skin within the target region of the electrode belt
* Unstable spine injury
* Body mass index of more than 50 kg/m2
* Incapacity to lie quietly for the examination
* Pacemaker, defibrillator or other active implant
* Reoperation before the examination at the third postoperative day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult inpatients undergoing elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in regional ventilation at the first postoperative day | baseline and 1. postoperative day
  Regional ventilation is measured by pulmonary electrical impedance tomography. The change in the calculated 'Center of Ventilation' in the sagittal direction is used for the primary outcome measure. Power calculation accounts for the use of two time points for the primary outcome measure.
Change from baseline in regional ventilation at the third postoperative day | baseline and 3. postoperative day
  Regional ventilation is measured by pulmonary electrical impedance tomography. The change in the calculated 'Center of Ventilation' in the sagittal direction is used for the primary outcome measure. Power calculation accounts for the use of two time points for the primary outcome measure.

SECONDARY OUTCOMES:
Change in forced vital capacity (FVC) | baseline, 1. and 3. postoperative day
  Measured by spirometry. The best value of three attempts is used.

OTHER OUTCOMES:
Change in forced expiratory volume in one second (FEV1) | baseline, 1. and 3. postoperative day
  Measured by spirometry. The best value of three attempts is used.
Change in peripheral oxygen saturation | baseline, 1. and 3. postoperative day
  Measured by pulse oximetry
Change in pain score | baseline, 1. and 3. postoperative day
  Measured by visual analogue scale
Change in respiratory rate | baseline, 1. and 3. postoperative day
  Measured by electric impedance tomography
pulmonary complications | baseline, 1., 3. and 7. postoperative day or at discharge
  Defined as pulmonary infection, pleural effusion, atelectasis, pneumothorax, bronchospasm, aspiration pneumonitis or respiratory insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Markus Kredel, PD. Dr. med, Principal Investigator — University of Würzburg, Department of Anaesthesia and Critical Care
Locations (1):
- University of Würzburg, Würzburg, Germany

REFERENCES:
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Mazo V, Sabate S, Canet J, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P. Prospective external validation of a predictive score for postoperative pulmonary complications. Anesthesiology. 2014 Aug;121(2):219-31. doi: 10.1097/ALN.0000000000000334. PMID 24901240
- [Background] Karayiannakis AJ, Makri GG, Mantzioka A, Karousos D, Karatzas G. Postoperative pulmonary function after laparoscopic and open cholecystectomy. Br J Anaesth. 1996 Oct;77(4):448-52. doi: 10.1093/bja/77.4.448. PMID 8942326
- [Background] Guizilini S, Bolzan DW, Faresin SM, Alves FA, Gomes WJ. Ministernotomy in myocardial revascularization preserves postoperative pulmonary function. Arq Bras Cardiol. 2010 Oct;95(5):587-93. doi: 10.1590/s0066-782x2010005000137. Epub 2010 Oct 15. English, Portuguese. PMID 20963310
- [Background] Davoudi M, Farhanchi A, Moradi A, Bakhshaei MH, Safarpour G. The Effect of Low Tidal Volume Ventilation during Cardiopulmonary Bypass on Postoperative Pulmonary Function. J Tehran Heart Cent. 2010 Summer;5(3):128-31. Epub 2010 Aug 31. PMID 23074580
- [Background] Leonhardt S, Lachmann B. Electrical impedance tomography: the holy grail of ventilation and perfusion monitoring? Intensive Care Med. 2012 Dec;38(12):1917-29. doi: 10.1007/s00134-012-2684-z. Epub 2012 Sep 20. PMID 22992946
- [Background] Radke OC, Schneider T, Heller AR, Koch T. Spontaneous breathing during general anesthesia prevents the ventral redistribution of ventilation as detected by electrical impedance tomography: a randomized trial. Anesthesiology. 2012 Jun;116(6):1227-34. doi: 10.1097/ALN.0b013e318256ee08. PMID 22531334
- [Background] Karsten J, Heinze H, Meier T. Impact of PEEP during laparoscopic surgery on early postoperative ventilation distribution visualized by electrical impedance tomography. Minerva Anestesiol. 2014 Feb;80(2):158-66. Epub 2013 Jul 23. PMID 23877309
- [Background] Frerichs I, Hahn G, Golisch W, Kurpitz M, Burchardi H, Hellige G. Monitoring perioperative changes in distribution of pulmonary ventilation by functional electrical impedance tomography. Acta Anaesthesiol Scand. 1998 Jul;42(6):721-6. doi: 10.1111/j.1399-6576.1998.tb05308.x. PMID 9689281
- [Derived] Bauer M, Opitz A, Filser J, Jansen H, Meffert RH, Germer CT, Roewer N, Muellenbach RM, Kredel M. Perioperative redistribution of regional ventilation and pulmonary function: a prospective observational study in two cohorts of patients at risk for postoperative pulmonary complications. BMC Anesthesiol. 2019 Jul 27;19(1):132. doi: 10.1186/s12871-019-0805-8. PMID 31351452